CLINICAL TRIAL: NCT04448561
Title: A Phase 1 Randomized, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Doses of ASP8062 With a Single Dose of Morphine in Recreational Opioid Using Participants
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Doses of ASP8062 With a Single Dose of Morphine in Recreational Opioid Using Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8062-CL-2002; UG3DA051392 (NIH)
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Results first posted 2021-09-29 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder; pharmacokinetic; ASP8062; morphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP8062 in combination with morphine (Experimental): Participants received ASP8062 tablet, orally once daily on days 1 through 10. On day 10, participants also received morphine tablet as single oral dose immediately after the ASP8062 dose.
  Interventions: Drug: ASP8082; Drug: morphine
- Placebo in combination with morphine (Placebo Comparator): Participants received ASP8062 matching placebo tablet, orally once daily on days 1 through 10. On day 10, participants also received morphine tablet as single oral dose immediately after the ASP8062 matching placebo dose.
  Interventions: Drug: morphine; Drug: Placebo

INTERVENTIONS:
Drug: ASP8082 — oral
  Arms: ASP8062 in combination with morphine
Drug: morphine — oral
Drug: Placebo — oral
  Arms: Placebo in combination with morphine

SUMMARY:
The primary purpose of this study was to assess the safety and tolerability of multiple doses of ASP8062 or placebo alone and in combination with a single dose of morphine.

This study also assessed the potential for pharmacokinetic interaction between ASP8062 and morphine.

DETAILED DESCRIPTION:
Participants were screened for up to 28 days prior to first investigational product administration. Eligible participants were admitted to the clinical unit on day -1 and were residential for a single period of 17 days/16 nights.

Participants were discharged from the clinical unit on day 16 on the condition that all required assessments had been performed and that there were no medical reasons for a longer stay in the clinical unit.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a recreational opioid user who has used opioids for nontherapeutic (recreational) purposes on at least 10 occasions within their lifetime, with at least 1 opioid use in the last 90 days.
* Participant has a body mass index (BMI) range of 18 to 36 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 28 days after final investigational product (IP) administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 28 days after final IP administration.
* Female participant must not donate ova starting at first dose of IP and throughout the study period and for 28 days after final IP administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for 90 days after final IP administration.
* Male participant must not donate sperm during the treatment period and for 90 days after final IP administration.
* Male participant with a pregnant partner(s) must agree to remain abstinent or use a condom with spermicide for the duration of the pregnancy throughout the study period and for 90 days after final IP administration.
* Participant agrees to not participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any condition which makes the participant unsuitable for study participation.
* Female participant who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Participant has a known or suspected hypersensitivity to ASP8062 or morphine and/or other opioids, or any components of the formulations used.
* Participant has had previous exposure with ASP8062.
* Participant has any of the liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase and total bilirubin [TBL]) ≥ 1.5 × upper limit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Participant has any clinically significant history of allergic conditions (including drug allergies, asthma or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to first IP administration.
* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal and/or other major disease or malignancy with exception of history of cholecystectomy.
* Participant has a history of moderate or severe use disorder for any substance other than caffeine or tobacco (based on the Diagnostic and Statistical Manual of Mental Disorders, edition 5 (DSM-5) criteria).
* Participant has a history or presence of any clinically significant psychiatric disorders such as, bipolar 1, schizophrenia, schizoaffective disorder or major depressive disorders.
* Participant has had recent suicidal ideation within the last 12 months or participant who is at significant risk to commit suicide using the Baseline/Screening Columbia-suicide severity rating scale (C-SSRS) at screening and the Since Last Visit C-SSRS on day -1.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Participant has any clinically significant abnormality following an investigator's review of the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -1.
* Participant has a mean pulse < 50 or > 90 bpm; mean systolic blood pressure > 150 mmHg; mean diastolic blood pressure > 95 mmHg (measurements taken in duplicate after participant has been resting in the supine position for at least 5 minutes) on day -1. If the mean blood pressure exceeds the limits above, 1 additional duplicate may be taken.
* Participant has a mean corrected QT interval using Fridericia's formula (QTcF) of > 450 msec (for male participants) and > 470 msec (for female participants) on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Participant has a positive test for amphetamines, barbiturates, benzodiazepines, cocaine, phencyclidine, alcohol and/or opiates on day -1. Positive tetrahydrocannabinol is not exclusionary and a cannabis intoxication evaluation will be performed. Participant may be reconsidered.
* Participant has used any prescribed or nonprescribed drugs (including vitamins and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to first IP administration, except for occasional use of acetaminophen (up to 2 g/day), topical dermatological products, including corticosteroid products, hormonal contraceptives and hormone replacement therapy (HRT).
* Participant must be willing to abstain from smoking (including use of tobacco-containing products and nicotine or nicotine-containing products [e.g., electronic vapes]) from at least 1 hour predose through at least 8 hours postdose on days 9 and 10.
* Participant has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Participant has had significant blood loss, donated approximately 500 mL of whole blood (excluding plasma donation) within 56 days prior to screening or donated plasma within 7 days prior to day -1.
* Participant has a positive serology test for hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at screening.
* Participant has loss of ability to freely provide consent through imprisonment or involuntary incarceration for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
* Participant is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/8062-CL-2002/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14566&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were recreational opioid users were enrolled in this study. Participants were enrolled in one site in the United States.
Pre-assignment Details: Eligible participants were randomized to ASP8062 or placebo using 2:1 ratio according to the randomization schedule. Participants who met the inclusion criteria and met none of the exclusion criteria were enrolled. A total of 54 participants were screened, out of which 30 participants failed screening.
Period: Overall Study
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine
Started | 16 | 8
Completed | 15 | 8
Not Completed | 1 | 0
Not completed — Noncompliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized: All participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (8.9) | 35.4 (10.4) | 32.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 12 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 5 | 16
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Blood Oxygen Saturation (SpO2) [Mean (Standard Deviation); unit: Percentage of oxygen saturation] — The SpO2 was measured using a pulse oximeter placed on the participant's fingertip. Baseline for SpO2 measurement was the last non-missing observation prior to first administration of ASP8062 or placebo.
  Percentage of oxygen saturation | 98.1 (1.0) | 98.8 (0.9) | 98.3 (1.0)
End Tidal Carbon Dioxide (CO2) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] — End tidal CO2 measurement was obtained per participant utilizing a portable bedside capnography device. The baseline for end tidal CO2 measurement was day 9, prior to dosing with ASP8062 or placebo. Population: Safety Analysis Set (SAF) with baseline value taken at Day 9. SAF included all participants randomly assigned to ASP8062 or placebo and who took at least 1 dose of ASP8062 or placebo. One participant from arm ASP8062 discontinued from study on day 2.
  millimeter of mercury (mmHg)
    number analyzed (Participants) | 15 | 8 | 23
    (all) | 37.1 (3.1) | 36.3 (2.2) | 36.8 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety was assessed by adverse events (AEs), which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study drug or was clinically significant. A Treatment emergent AE (TEAE) was defined as any AE that started or worsened after the first dose of study drug up to 30 days after the last dose of study drug. AEs were considered serious (SAEs) if the AE resulted in death, was life-threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly, or birth defect or required inpatient hospitalization or led to prolongation of hospitalization.
Time Frame: From first dose of study drug up to end of study visit (up to day 25)
Population: The analysis population was the SAF, which consisted of all participants randomly assigned to investigational product (ASP8062 or placebo) and who took at least 1 dose of investigational product (ASP8062 or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- ASP8062: Participants received ASP8062 tablet, orally once daily on days 1 through 9.
- ASP8062 in Combination With Morphine: Participants received ASP8062 tablet, orally once on day 10. On day 10, participants also received morphine tablet as single oral dose immediately after the ASP8062 dose.
- Placebo: Participants received ASP8062 matching placebo tablet, orally once daily on days 1 through 9.
- Placebo in Combination With Morphine: Participants received ASP8062 matching placebo tablet, orally once on day 10. On day 10, participants also received morphine tablet as single oral dose immediately after the ASP8062 matching placebo dose.
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 16 | 15 | 8 | 8
Participants
  TEAE | 7 | 11 | 3 | 7
  Drug-related TEAE | 6 | 11 | 3 | 7
  Serious TEAE | 0 | 0 | 0 | 0
  Drug-related serious TEAE | 0 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0
  Drug related TEAE leading to death | 0 | 0 | 0 | 0
  TEAE leading to withdrawal of treatment | 0 | 0 | 0 | 0
  Drug-related TEAE leading to withdrawal of treatment | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With At Least One Event of Suicidal Ideation And/or Suicidal Behavior as Assessed by The Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a clinician administered assessment tool that evaluates suicidal ideation and behavior. Number of participants with at least one affirmative response to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 5 items for suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide) were reported.
Time Frame: Up to day 25
Population: The analysis population was the SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 16 | 15 | 8 | 8
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at Predose
Description: The SpO2 was measured using a pulse oximeter placed on the participant's fingertip. Change from baseline in SpO2 was calculated as Day 9 minus Baseline for arms 'ASP8062' and 'Placebo', and Day 10 minus Baseline for arms 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine'. Baseline observation was last non-missing observation prior to first dose.
Time Frame: 'ASP8062' and 'Placebo': Baseline and predose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline and predose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
percentage of oxygen saturation | 0.4 (1.3) | 0.3 (1.2) | -0.5 (0.8) | -0.6 (1.3)

4. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 1 Hour Postdose
Description: as for outcome 3
Time Frame: 'ASP8062' and 'Placebo': Baseline and 1 hour postdose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline and 1 hour postdose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
percentage of oxygen saturation | 0.1 (1.4) | -0.7 (1.4) | -0.5 (1.4) | -1.4 (1.7)

5. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 2 Hour Postdose
Description: as for outcome 3
Time Frame: 'ASP8062' and 'Placebo': Baseline and 2 hour postdose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline and 2 hour postdose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
percentage of oxygen saturation | -0.1 (1.2) | -0.5 (1.6) | -0.9 (1.1) | -0.6 (0.9)

6. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 4 Hour Postdose
Description: as for outcome 3
Time Frame: 'ASP8062' and 'Placebo': Baseline and 4 hour postdose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline and 4 hour postdose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
percentage of oxygen saturation | 0.1 (1.5) | -0.2 (1.1) | -0.5 (1.1) | -1.0 (1.6)

7. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 8 Hour Postdose
Description: as for outcome 3
Time Frame: 'ASP8062' and 'Placebo': Baseline and 8 hour postdose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline and 8 hour postdose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
percentage of oxygen saturation | 0.0 (1.6) | -0.5 (2.3) | -1.1 (1.8) | -0.5 (1.6)

8. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 12 Hour Postdose
Description: as for outcome 3
Time Frame: 'ASP8062' and 'Placebo': Baseline and 12 hour postdose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline and 12 hour postdose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
percentage of oxygen saturation | -0.4 (1.6) | -0.5 (1.3) | -1.5 (1.8) | -1.3 (1.7)

9. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at Predose
Description: End tidal CO2 measurement was obtained per participant utilizing a portable bedside capnography device. Change from baseline in CO2 was calculated as Day 9 minus Baseline for arms 'ASP8062' and 'Placebo', and Day 10 minus Baseline (baseline observation was observation before first dose at Day 9) for arms 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine'.
Time Frame: 'ASP8062' and 'Placebo': Baseline and predose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline (observation taken at Day 9), and predose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
mmHg | NA (NA) — predose CO2 assessment was not performed for this group on Day 9. | -1.0 (2.4) | NA (NA) — predose CO2 assessment was not performed for this group on Day 9. | 0.5 (3.3)

10. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at 1 Hour Postdose
Description: as for outcome 9
Time Frame: 'ASP8062' and 'Placebo': Baseline and 1 hour postdose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline (observation taken at Day 9), and 1 hour postdose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
mmHg | -0.9 (2.4) | 0.7 (2.3) | -0.4 (4.4) | 2.5 (2.6)

11. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at 2 Hour Postdose
Description: as for outcome 9
Time Frame: 'ASP8062' and 'Placebo': Baseline and 2 hour postdose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline (observation taken at Day 9), and 2 hour postdose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
mmHg | -1.1 (2.5) | 2.5 (3.2) | -1.0 (1.9) | 4.1 (2.7)

12. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at 4 Hour Postdose
Description: as for outcome 9
Time Frame: 'ASP8062' and 'Placebo': Baseline and 4 hour postdose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline (observation taken at Day 9), and 4 hour postdose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
mmHg | -0.8 (1.7) | 1.0 (2.6) | 0.1 (2.5) | 3.3 (2.0)

13. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at 8 Hour Postdose
Description: as for outcome 9
Time Frame: 'ASP8062' and 'Placebo': Baseline and 8 hour postdose Day 9; 'ASP8062 in combination with morphine' and 'Placebo in combination with morphine': Baseline (observation taken at Day 9), and 8 hour postdose Day 10
Population: SAF population with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 15 | 8 | 8
mmHg | 0.2 (0.3) | 2.7 (3.3) | 2.1 (1.5) | 5.8 (1.7)

14. Secondary Outcome: Pharmacokinetics (PK) of ASP8062 in Plasma: Area Under the Concentration From Time of Dosing to 24 Hours (AUC24)
Description: AUC24 was recorded from the PK plasma samples collected. Samples for AUC24 were collected for arm 'ASP8062' at Day 9, and for arm 'ASP8062 in combination with morphine' at Day 10.
Time Frame: 'ASP8062': Predose, 0.25, 0.5, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 h postdose Day 9; 'ASP8062 in combination with morphine': Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144 h postdose Day 10
Population: The analysis population was Pharmacokinetic Analysis Set (PKAS) with available data at each time point. PKAS consisted of all participants who received at least 1 dose of ASP8062 for which concentration data were available to facilitate derivation of at least 1 pharmacokinetic parameter of ASP8062.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter(ng*h/mL)
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine
Number analyzed (Participants) | 15 | 15
nanogram*hour per milliliter(ng*h/mL) | 1640 (619) | 1640 (589)
Statistical Analysis 1: Comparison: ASP8062 vs ASP8062 in Combination With Morphine; Test type: Other; Geometric Least square (LS) mean ratio = 100.64, 90% CI 2-sided [98.37 to 102.96] — Assessment based on analysis of variance performed on natural log-transformed parameters with treatment as fixed effect and participant as random effect. Ratios and confidence limits: transformed back to raw scale and values expressed as percentages

15. Secondary Outcome: Pharmacokinetics (PK) of ASP8062 in Plasma: Maximum Plasma Concentration (Cmax)
Description: Cmax was recorded from the PK plasma samples collected. Samples for Cmax were collected for arm 'ASP8062' at Day 9, and for arm 'ASP8062 in combination with morphine' at Day 10.
Time Frame: 'ASP8062': Predose, 0.25, 0.5, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 h Day 9; 'ASP8062 in combination with morphine': Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144 h postdose Day 10
Population: The analysis population was PKAS with available data at each time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine
Number analyzed (Participants) | 15 | 15
nanogram per milliliter (ng/mL) | 124 (41.1) | 116 (31.8)
Statistical Analysis 1: Comparison: ASP8062 vs ASP8062 in Combination With Morphine; Test type: Other; Geometric LS mean ratio = 94.28, 90% CI 2-sided [89.29 to 99.54] — [estimate comment as in outcome 14, analysis 1]

16. Secondary Outcome: Pharmacokinetics (PK) of Morphine in Plasma: Area Under the Concentration From Time of Dosing Extrapolated to Time Infinity (AUCinf)
Description: AUCinf was recorded from the PK plasma samples collected.
Time Frame: Predose, 0.25, 0.5, 1.5, 2, 3, 4, 8, 12, 16, 24, 36, 48 h postdose Day 10
Population: The analysis population was PKAS with available data at each time point. Insufficient number of samples were available for calculation for AUCinf.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine
Number analyzed (Participants) | 3 | 3
ng*h/mL | 128 (43.5) | 166 (13.7)

17. Secondary Outcome: Pharmacokinetics (PK) of Morphine in Plasma: Area Under the Concentration Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast)
Description: AUClast was recorded from the PK plasma samples collected.
Time Frame: Predose, 0.25, 0.5, 1.5, 2, 3, 4, 8, 12, 16, 24, 36, 48 h postdose Day 10
Population: The analysis population was PKAS.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 8
ng*h/mL | 160 (39.8) | 158 (42.1)
Statistical Analysis 1: Comparison: ASP8062 in Combination With Morphine vs Placebo in Combination With Morphine; Test type: Other; Geometric LS mean ratio = 100.79, 90% CI 2-sided [83.35 to 121.88] — Assessment based on an analysis of variance performed on natural log-transformed parameters with treatment as a fixed effect. Ratios and confidence limits were transformed back to raw scale and values were expressed as percentages

18. Secondary Outcome: Pharmacokinetics (PK) of Morphine in Plasma: Cmax
Description: Cmax was recorded from the PK plasma samples collected.
Time Frame: Predose, 0.25, 0.5, 1.5, 2, 3, 4, 8, 12, 16, 24, 36, 48 h postdose Day 10
Population: The analysis population was PKAS.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 8
ng/mL | 41.3 (9.17) | 42.3 (15.6)
Statistical Analysis 1: Comparison: ASP8062 in Combination With Morphine vs Placebo in Combination With Morphine; Test type: Other; Geometric LS mean ratio = 100.58, 90% CI 2-sided [81.35 to 124.36] — [estimate comment as in outcome 17, analysis 1]

19. Secondary Outcome: Pharmacokinetics (PK) of Morphine-3β-D-glucuronide(M3G) (Morphine Metabolite) in Plasma: AUCinf
Description: AUCinf was recorded from the PK plasma samples collected.
Time Frame: Predose, 0.25, 0.5, 1.5, 2, 3, 4, 8, 12, 16, 24, 36, 48 h postdose Day 10
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine
Number analyzed (Participants) | 7 | 6
ng*h/mL | 5720 (980) | 6580 (702)

20. Secondary Outcome: Pharmacokinetics (PK) of Morphine-3β-D-glucuronide (M3G) (Morphine Metabolite) in Plasma: AUClast
Description: AUClast was recorded from the PK plasma samples collected.
Time Frame: Predose, 0.25, 0.5, 1.5, 2, 3, 4, 8, 12, 16, 24, 36, 48 h postdose Day 10
Population: The analysis population was PKAS.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 8
ng*h/mL | 5340 (887) | 5960 (703)
Statistical Analysis 1: Comparison: ASP8062 in Combination With Morphine vs Placebo in Combination With Morphine; Test type: Other; Geometric LS mean ratio = 89.08, 90% CI 2-sided [79.58 to 99.71] — [estimate comment as in outcome 17, analysis 1]

21. Secondary Outcome: Pharmacokinetics (PK) of Morphine-3β-D-glucuronide (M3G) (Morphine Metabolite) in Plasma: Cmax
Description: Cmax was recorded from the PK plasma samples collected.
Time Frame: Predose, 0.25, 0.5, 1.5, 2, 3, 4, 8, 12, 16, 24, 36, 48 h postdose Day 10
Population: The analysis population was PKAS.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ASP8062 in Combination With Morphine: Participants received ASP8062 tablet, orally once day 10. On day 10, participants also received morphine tablet as single oral dose immediately after the ASP8062 dose.
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 8
ng/mL | 933 (189) | 967 (176)
Statistical Analysis 1: Comparison: ASP8062 in Combination With Morphine vs Placebo in Combination With Morphine; Test type: Other; Geometric LS mean ratio = 96.11, 90% CI 2-sided [83.03 to 111.25] — Assessment based on an analysis of variance performed on natural log-transformed parameters with treatment as a fixed effect. Ratios and confidence limits are transformed back to raw scale and values are expressed as percentages

22. Secondary Outcome: Pharmacokinetics (PK) of Morphine-6β-D-glucuronide (M6G) (Morphine Metabolite) in Plasma: AUCinf
Description: AUCinf was recorded from the PK plasma samples collected.
Time Frame: Predose, 0.25, 0.5, 1.5, 2, 3, 4, 8, 12, 16, 24, 36, 48 h postdose Day 10
Population: The analysis population was the PKAS with available at each time point. The analysis population was PKAS with available data at each time point. Insufficient number of samples were available for calculation for AUCinf.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine
Number analyzed (Participants) | 5 | 5
ng*h/mL | 821 (138) | 1100 (212)

23. Secondary Outcome: Pharmacokinetics (PK) of Morphine-6β-D-glucuronide (M6G) (Morphine Metabolite) in Plasma: AUClast
Description: AUClast was recorded from the PK plasma samples collected.
Time Frame: Predose, 0.25, 0.5, 1.5, 2, 3, 4, 8, 12, 16, 24, 36, 48 h postdose Day 10
Population: The analysis population was the PKAS.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ASP8062 in Combination With Morphine | Placebo in Combination With Morphine
Number analyzed (Participants) | 15 | 8
ng*h/mL | 871 (161) | 1000 (165)
Statistical Analysis 1: Comparison: ASP8062 in Combination With Morphine vs Placebo in Combination With Morphine; Test type: Other; Geometric LS mean ratio = 86.54, 90% CI 2-sided [76.01 to 98.52] — [estimate comment as in outcome 21, analysis 1]

24. Secondary Outcome: Pharmacokinetics (PK) of Morphine-6β-D-glucuronide (M6G) (Morphine Metabolite) in Plasma: Cmax
Description: Cmax was recorded from the PK plasma samples collected.
Time Frame: Predose, 0.25, 0.5, 1.5, 2, 3, 4, 8, 12, 16, 24, 36, 48 h postdose Day 10
Population: The analysis population was the PKAS.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Placebo Combination With Morphine: Participants received ASP8062 matching placebo tablet, orally once on day 10. On day 10, participants also received morphine tablet as single oral dose immediately after the ASP8062 matching placebo dose.
Arm/Group | ASP8062 in Combination With Morphine | Placebo Combination With Morphine
Number analyzed (Participants) | 15 | 8
ng/mL | 184 (37.6) | 192 (30.9)
Statistical Analysis 1: Comparison: ASP8062 in Combination With Morphine vs Placebo Combination With Morphine; Test type: Other; Geometric LS mean ratio = 95.10, 90% CI 2-sided [82.52 to 109.60] — [estimate comment as in outcome 17, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study visit (up to day 25)
Groups:
- Placebo: Participants received ASP8062 matching placebo tablet, orally once daily on days 1 through 9. On day 10, participants also received morphine tablet as single oral dose immediately after the ASP8062 matching placebo dose.
Arm/Group | ASP8062 | ASP8062 in Combination With Morphine | Placebo | Placebo in Combination With Morphine
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/16 | 11/15 | 3/8 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP8062 (N=16) | ASP8062 in Combination With Morphine (N=15) | Placebo (N=8) | Placebo in Combination With Morphine (N=8)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (3)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling of relaxation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (3) | 2 (2) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 1 (1) | 5 (5) | 0 (0) | 4 (4)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT04448561/Prot_SAP_000.pdf